CLINICAL TRIAL: NCT01482117
Title: Randomized, Open-label, Crossover Study to Evaluate the Effect of Genetic Polymorphism on Pharmacokinetic & Pharmacodynamic Interactions of Clopidogrel and Cilostazol in Korean Healthy Adult Volunteers
Brief Title: The Effect of Genetic Polymorphism on Interactions of Clopidogrel and Cilostazol in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jae-Gook Shin, Department of Pharmacology and Pharmacogenomics Research Center, Inje University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-105
Record Dates: First submitted 2011-11-26; First posted 2011-11-30 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Interaction
Keywords: CYP2C19; CYP3A5; Clopidogrel; Cilostazol; Healthy
MeSH Terms: interventions — Clopidogrel; Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clopidogrel (Active Comparator): single oral administration of 300mg of clopidogrel
  Interventions: Drug: Clopidogrel; Drug: Cilostazol; Drug: Clopidogrel/Cilostazol
- Cilostarole (Active Comparator): single oral administration of 100mg of cilostazole
  Interventions: Drug: Clopidogrel; Drug: Cilostazol; Drug: Clopidogrel/Cilostazol
- Clopidogrel/Cilostazol (Active Comparator): single oral administration of 300mg clopidogrel and 100mg cilostazol
  Interventions: Drug: Clopidogrel; Drug: Cilostazol; Drug: Clopidogrel/Cilostazol

INTERVENTIONS:
Drug: Clopidogrel — single oral administration of 300mg of clopidogrel
  Other Names: Plavix
Drug: Cilostazol — single oral administration of 100mg cilostazol
  Other Names: Pletaal
Drug: Clopidogrel/Cilostazol — single oral administration of 300mg clopidogrel and 100mg cilostazol
  Other Names: Plavix/Pletaal

SUMMARY:
The aim of this study is to investigate the effects of genetic polymorphisms on pharmacokinetic and pharmacodynamic interactions of clopidogrel and cilostazol in Korean healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject whose CYP2C19 genotype was determined

Exclusion Criteria:

* Subject who has abnormal laboratory test results

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Maximum concentration(Cmax), Area under the concentration(AUC), Inhibition of platelet aggregation(IPA) | up to 24 hours
  9 or 11 point blood sampling according to the interventions

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Gook Shin, MD, PhD, Principal Investigator — Inje University